CLINICAL TRIAL: NCT04126200
Title: A Phase I/II, Randomized, Open-label Platform Study Utilizing a Master Protocol to Study Belantamab Mafodotin (GSK2857916) as Monotherapy and in Combination With Anti-Cancer Treatments in Participants With Relapsed/Refractory Multiple Myeloma (RRMM) - DREAMM 5
Brief Title: Platform Study of Belantamab Mafodotin as Monotherapy and in Combination With Anti-cancer Treatments in Participants With Relapsed/Refractory Multiple Myeloma (RRMM)
Acronym: DREAMM5
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 208887
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Belantamab mafodotin; GSK2857916; GSK3174998; Feladilimab; Nirogacestat; Dostarlimab; Isatuximab; Lenalidomide; Dexamethasone; Pomalidomide; Platform study; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; nirogacestat; dostarlimab; isatuximab; Lenalidomide; Dexamethasone; pomalidomide

STUDY DESIGN:
Intervention Model Description: There will be a dose exploration (DE) phase which will evaluate the safety and tolerability profile of belantamab mafodotin when administered in combination with other anti-cancer treatments. A recommended Phase 2 dose (RP2D) for each combination treatment will be identified based on the safety and preliminary efficacy in DE. This will be followed by a cohort expansion (CE) phase which will evaluate the clinical activity of the combination treatment in comparison to belantamab mafodotin monotherapy in additional participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (17):
- Belantamab mafodotin+GSK3174998 dose exploration (Sub-study 1) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: GSK3174998
- Belantamab mafodotin+feladilimab dose exploration (Sub-study 2) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Feladilimab
- Belantamab mafodotin+nirogacestat dose exploration(Sub-study 3) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat
- Belantamab mafodotin+dostarlimab dose exploration(Sub-study 4) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dostarlimab
- Belantamab mafodotin+isatuximab dose exploration (Sub-study 5) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Isatuximab
- Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 6) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Lenalidomide; Drug: Dexamethasone
- Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone dose exploration (Sub-study 7) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Dexamethasone; Drug: Pomalidomide
- Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 8) (Experimental): This cohort will enroll Northeast Asian participants.
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Lenalidomide; Drug: Dexamethasone
- Belantamab mafodotin monotherapy cohort expansion (Active Comparator)
  Interventions: Drug: Belantamab mafodotin
- Belantamab mafodotin+GSK3174998 cohort expansion (Sub-study 1) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: GSK3174998
- Belantamab mafodotin+ feladilimab cohort expansion (Sub-study 2) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Feladilimab
- Belantamab mafodotin+ nirogacestat cohort expansion (Sub-study 3) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat
- Belantamab mafodotin+ dostarlimab cohort expansion (Sub-study 4) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Dostarlimab
- Belantamab mafodotin+ isatuximab cohort expansion (Sub-study 5) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Isatuximab
- Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 6) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Lenalidomide; Drug: Dexamethasone
- Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone cohort expansion (Sub-study 7) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Dexamethasone; Drug: Pomalidomide
- Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 8) (Experimental): This cohort will enroll Northeast Asian participants.
  Interventions: Drug: Belantamab mafodotin; Drug: Nirogacestat; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
Drug: GSK3174998 — GSK3174998 will be administered.
  Arms: Belantamab mafodotin+GSK3174998 cohort expansion (Sub-study 1); Belantamab mafodotin+GSK3174998 dose exploration (Sub-study 1)
Drug: Feladilimab — feladilimab will be administered.
  Arms: Belantamab mafodotin+ feladilimab cohort expansion (Sub-study 2); Belantamab mafodotin+feladilimab dose exploration (Sub-study 2)
Drug: Nirogacestat — Nirogacestat will be administered.
  Arms: Belantamab mafodotin+ nirogacestat cohort expansion (Sub-study 3); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 8); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 8); Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone cohort expansion (Sub-study 7); Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone dose exploration (Sub-study 7); Belantamab mafodotin+nirogacestat dose exploration(Sub-study 3)
Drug: Dostarlimab — Dostarlimab will be administered.
  Arms: Belantamab mafodotin+ dostarlimab cohort expansion (Sub-study 4); Belantamab mafodotin+dostarlimab dose exploration(Sub-study 4)
Drug: Isatuximab — Isatuximab will be administered.
  Arms: Belantamab mafodotin+ isatuximab cohort expansion (Sub-study 5); Belantamab mafodotin+isatuximab dose exploration (Sub-study 5)
Drug: Lenalidomide — Lenalidomide will be administered.
  Arms: Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 8); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 8)
Drug: Dexamethasone — Dexamethasone will be administered.
  Arms: Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone cohort expansion (Sub-study 8); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 6); Belantamab mafodotin+ nirogacestat+ lenalidomide+ dexamethasone dose exploration (Sub-study 8); Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone cohort expansion (Sub-study 7); Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone dose exploration (Sub-study 7)
Drug: Pomalidomide — Pomalidomide will be administered.
  Arms: Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone cohort expansion (Sub-study 7); Belantamab mafodotin+ nirogacestat+ pomalidomide + dexamethasone dose exploration (Sub-study 7)

SUMMARY:
B-cell maturation antigen (BCMA) is a target present on tumor cells in participants with multiple myeloma. Belantamab mafodotin (GSK2857916); is an antibody-drug conjugate (ADC) containing humanized anti-BCMA monoclonal antibody (mAb). This is a phase I/II, randomized, open-label, platform study designed to evaluate the effects of belantamab mafodotin in combination with other anti-cancer drugs in participants with relapsed/refractory multiple myeloma. The Platform design incorporates a single master protocol, where multiple treatment combinations, as sub-studies, will be evaluated simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older, at the time of signing the informed consent.
* Participants must have histologically or cytologically confirmed diagnosis of Multiple Myeloma (MM), as defined by the IMWG.
* Participants having at least 3 prior lines of prior anti-myeloma treatments including an immunomodulating agent (IMID) a proteasome inhibitor (PI) and an anti-CD38 monoclonal antibody.
* Participants with a history of autologous stem cell transplant are eligible for study participation when, transplant was >100 days prior to study enrolment and with no active infection(s).
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, unless ECOG less than equal to (<=)2 is due solely to skeletal complications and/or skeletal pain due to MM.
* Participants with measurable disease defined as at least one of the following: Serum M-protein greater than equal to (>=)0.5 gram per deciliter (>=5 gram per liter) or Urine M-protein >=200 milligrams (mg) per 24 hours or Serum free light chain (FLC) assay: Involved FLC level >=10 mg per deciliter (>=100 mg per Liter) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participants who have tested positive for Hepatitis B core antibody (HBcAb) can be enrolled if the following criteria are met: Serology result HBcAb+, Hepatitis B surface antigen (HBsAg)-; HBV deoxyribonucleic acid (DNA) undetectable during screening.
* Participants who are currently receiving physiological doses oral steroids (<10 mg/day), inhaled steroids or ophthalmalogical steroids.

Inclusion Criteria Specific to Sub-study 6,7, and 8:

* Participants with contraception requirements specific to Sub-study 6, 7, and 8 respectively.
* Participants with platelets value for Adequate Organ System Function is ≥75 × 10^9/L.

Inclusion Criteria Specific to Sub-study 8:

- In Japan, participants should reside in Japan and be Japanese as defined by having all biological Japanese grandparents. Similarly, in China, subjects should reside in China and be Chinese as defined by having all biological Chinese grandparents.

Exclusion Criteria:

* Participants with current corneal epithelial disease except mild punctate keratopathy.
* Participants with evidence of cardiovascular risk.
* Participants with known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to belantamab mafodotin or any of the components of the study treatment. History of severe hypersensitivity to other mAb.
* Participants with active infection requiring antibiotic, antiviral, or antifungal treatment.
* Participants with other monoclonal antibodies within 30 days or systemic anti-myeloma therapy within <14 days.
* Participants with prior radiotherapy within 2 weeks of start of study therapy.
* Participants with prior allogeneic transplant are prohibited.
* Participants who have received prior Chimeric Antigen T cell therapy (CAR-T) therapy with lymphodepletion with chemotherapy within 3 months of screening.
* Participants with any major surgery (other than bone-stabilizing surgery) within the last 30 days.
* Participants with prior treatment with an investigational agent within 14 days or 5 half-lives of receiving the first dose of study drugs, whichever is shorter.
* Participants with >=grade 3 toxicity considered related to prior check-point inhibitors and that led to treatment discontinuation.
* Participants who have received transfusion of blood products within 2 weeks before the first dose of study drug.
* Participants must not receive live attenuated vaccines within 30 days prior to first dose of study treatment or whilst receiving belantamab mafodotin +- partner agent in any sub-study arm of the platform trial and for at least 70 days following last study treatment.
* Participants with presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM.
* Participants with known human immunodeficiency virus (HIV) infection, unless the participant can meet all criteria: a) established anti-retroviral therapy for at least 4 weeks and HIV viral load<400 copies/milliliter (mL) b) cluster of differentiation 4 plus (CD4+) T-cell (CD4+) counts >= 350 cells/microliter (µL) c) No history of Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months in which case the participant would be eligible for CE Phase only.

For participants receiving nirogacestat, HIV drugs that are strong Cytochrome P450 3A4 (CYP3A4) inhibitors are prohibited. HIV drugs that are moderate CYP3A4 inhibitors, while permitted, should be co-administered with caution and must be accompanied by nirogacestat dose modifications.

Additional Exclusion Criteria for Sub-study 1 and 2:

* Participants with autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years.
* Exclusion for a recent (within the past 6 months) history of symptomatic pericarditis.

Additional Exclusion Criteria for Sub-study 3, 6, 7, and 8:

* Participants with uncontrolled small and/or large intestinal disease.
* Participants with uncontrolled skin disease.
* Participants with any condition causing hypophosphatemia, hypokalemia or hypomagnesemia which is refractory to electrolyte replacement.
* Participants with previous administration of a gamma secretase inhibitor.
* Participants with concomitant administration of a strong CYP3A4 inhibitor or inducer.

Additional Exclusion Criteria for Sub-study 4:

* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Participants who have received prior therapy with an anti-programmed death-1 (anti-PD-1), anti-PD-1-ligand-1 (anti-PD-L1), or anti-PD-1 ligand-2 (anti-PD-L2) agent.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. Use of inhaled steroids, local injection of steroids, and steroid eye drops are allowed.

Additional Exclusion Criteria for Sub-study 5:

* Participants with Severe hypersensitivity to Isatuximab-irfc or to any of its excipients.
* Participants with prior treatment with other anti-CD38 monoclonal antibody within 6 months of the first dose of study drug treatment.
* Participants with known intolerance or hypersensitivity to infused proteins products, sucrose, histidine, and polysorbate 80.

Additional Exclusion Criteria for Sub-study 6, 7, and 8:

* Participants with active or history of venous thromboembolism within the past 3 months.
* Participants with evidence of active mucosal or internal bleeding.
* Participants with contraindications to or are unwilling to undergo protocol-required anti-thrombotic prophylaxis or unable to tolerate antithrombolitic prophalaxis.

Additional Exclusion Criteria for Sub-study 6 and 8:

- Participants who discontinued prior treatment with lenalidomide due to intolerable adverse events.

Additional Exclusion Criteria for Sub-study 7:

- Participants who discontinued prior treatment with pomalidomide due to intolerable adverse events.

Additional Exclusion Criteria for Sub-study 8:

* Pregnant or lactating female or female who are interrupting lactation.
* Previously diagnosed with interstitial lung disease or current complication of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
DE Phase: Number of participants achieving dose limiting toxicities (DLT) | Up to 12 months
  An event is considered to be a DLT if the event occurs within the first 28 days of treatment and meets protocol defined DLT criteria.
DE Phase: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 12 months
  AEs and SAEs will be collected.
DE Phase: Number of participants with clinically significant changes in hematology, clinical chemistry and urinalysis lab parameters | Up to 12 months
  Blood and urine samples will be collected to evaluate hematology, clinical chemistry and urinalysis lab parameters.
CE Phase: Number of participants achieving Overall Response Rate (ORR) | Up to 36 months
  ORR is defined as the percentage of participants with a Partial response (PR) or better, according to the International Myeloma Working Group (IMWG) Response Criteria.

SECONDARY OUTCOMES:
DE Phase: Number of participants achieving ORR | Up to 12 months
  ORR is defined as the percentage of participants with PR or better, according to the IMWG Response Criteria.
CE Phase: Number of participants achieving Clinical Benefit Rate (CBR) | Up to 36 months
  CBR is defined as the percentage of participants with a minimal response (MR) or better, according to IMWG response criteria.
DE Phase: Number of participants achieving Partial Response (PR) | Up to 12 months
  Number of participants with PR according to IMWG criteria will be analyzed.
CE Phase: Number of participants achieving PR | Up to 36 months
  Number of participants with PR according to IMWG criteria will be analyzed.
DE Phase: Number of participants achieving Very Good Partial Response (VGPR) | Up to 12 months
  Number of participants with VGPR according to IMWG criteria will be analyzed.
CE Phase: Number of participants achieving VGPR | Up to 36 months
  Number of participants with VGPR according to IMWG criteria will be analyzed.
DE Phase: Number of participants achieving Complete Response (CR) | Up to 12 months
  Participants with CR according to IMWG criteria will be analyzed.
CE Phase: Number of participants achieving CR | Up to 36 months
  Participants with CR according to IMWG criteria will be analyzed.
DE Phase: Number of participants achieving stringent Complete Response (sCR) | Up to 12 months
  Participants with sCR according to IMWG criteria will be analyzed.
CE Phase: Number of participants achieving sCR | Up to 36 months
  Participants with sCR according to IMWG criteria will be analyzed.
DE Phase: Belantamab mafodotin concentrations when administered in combination with anti-cancer treatments | Up to 12 months
  Blood samples will be collected for concentrations of belantamab mafodotin.
CE Phase: Belantamab mafodotin concentrations when administered in combination with anti-cancer treatments | Up to 36 months
  Blood samples will be collected for concentrations of belantamab mafodotin.
DE Phase: GSK3174998 concentration when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples will be collected for concentrations of GSK3174998.
CE Phase: GSK3174998 concentration when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples will be collected for concentrations of GSK3174998.
DE Phase: Feladilimab concentration when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples will be collected for concentrations of feladilimab.
CE Phase: Feladilimab concentration when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples will be collected for concentrations of feladilimab.
DE Phase: Nirogacestat concentration when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples will be collected for concentrations of nirogacestat.
CE Phase: Nirogacestat concentration when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples will be collected for concentrations of nirogacestat.
DE Phase: Dostarlimab concentration when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples will be collected for concentrations of dostarlimab.
CE Phase: Dostarlimab concentration when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples will be collected for concentrations of dostarlimab.
DE Phase: Isatuximab concentration when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples will be collected for concentrations of isatuximab.
CE Phase: Isatuximab concentration when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples will be collected for concentrations of isatuximab.
DE Phase: Concentration of anti-drug antibodies (ADAs) against belantamab mafodotin when administered in combination with anti-cancer treatments | Up to 12 months
  Blood samples for concentrations for ADAs will be collected.
CE Phase: Concentration of ADAs against belantamab mafodotin when administered in combination with anti-cancer treatments | Up to 36 months
  Blood samples for concentrations for ADAs will be collected.
DE Phase: Concentration of ADAs against GSK3174998 when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples for concentrations for ADAs will be collected.
CE Phase: Concentration of ADAs against GSK3174998 when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples for concentrations for ADAs will be collected.
DE Phase: Concentration of ADAs against feladilimab when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples for concentrations for ADAs will be collected.
CE Phase: Concentration of ADAs against feladilimab when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples for concentrations for ADAs will be collected.
DE Phase: Concentration of ADAs against dostarlimab when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples for concentrations for ADAs will be collected.
CE Phase: Concentration of ADAs against dostarlimab when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples for concentrations for ADAs will be collected.
DE Phase: Concentration of ADAs against isatuximab when administered in combination with belantamab mafodotin | Up to 12 months
  Blood samples for concentrations for ADAs will be collected.
CE Phase: Concentration of ADAs against isatuximab when administered in combination with belantamab mafodotin | Up to 36 months
  Blood samples for concentrations for ADAs will be collected.
DE Phase: Number of participants with adverse events of special interest (AESI) for belantamab mafodotin | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for belantamab mafodotin | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with AESI for GSK3174998 | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for GSK3174998 | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with AESI for Feladilimab | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for Feladilimab | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with AESI for Nirogacestat | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for Nirogacestat | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with AESI for Dostarlimab | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for Dostarlimab | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with AESI for Isatuximab | Up to 12 months
  AESIs will be collected.
CE Phase: Number of participants with AESI for Isatuximab | Up to 36 months
  AESIs will be collected.
DE Phase: Number of participants with abnormal ocular findings on ophthalmic examination | Up to 12 months
  Ophthalmic examination will assess abnormal findings.
CE Phase: Number of participants with abnormal ocular findings on ophthalmic examination | Up to 36 months
  Ophthalmic examination will assess abnormal findings.
CE Phase: Number of participants achieving Progression-free survival (PFS) | Up to 36 months
  PFS is defined as the time from randomization until the earliest date of confirmed progressive disease (PD) per IMWG, or death due to any cause.
CE Phase: Duration of response (DoR) | Up to 36 months
  DoR is defined as the time from first documented evidence or PR or better until progressive disease per IMWG or death due to progressive disease among participants who achieve confirmed partial response or better.
CE Phase: Time to response (TTR) | Up to 36 months
  TTR is defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (confirmed PR or better).
CE Phase: Number of participants achieving Overall survival (OS) | Up to 36 months
  OS is defined as the time from randomization until death due to any cause.
CE Phase: Number of participants with AEs and SAEs | Up to 36 months
  AEs and SAEs will be collected.
CE Phase: Number of participants with AEs leading to discontinuation | Up to 36 months
  Number of participants with AEs leading to discontinuation will be evaluated.
CE Phase: Number of participants with dose reduction or delay | Up to 36 months
  Number of participants with dose reduction or delay will be evaluated.
CE Phase: Number of participants with clinically significant changes in hematology, clinical chemistry and urinalysis lab parameters | Up to 36 months
  Blood and urine samples will be collected to evaluate hematology, clinical chemistry and urinalysis lab parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (5):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Madison, Wisconsin
- Australia (2):
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Brazil (3):
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
- France (2):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Villejuif
- Germany (4):
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Kiel
  - GSK Investigational Site, Leipzig
- GSK Investigational Site, Athens, Greece
- GSK Investigational Site, Mexico City, Mexico
- Netherlands (2):
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Utrecht
- GSK Investigational Site, Oslo, Norway
- Poland (4):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
- GSK Investigational Site, Moscow, Russia
- South Korea (3):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
- Sweden (2):
  - GSK Investigational Site, Falun
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hosoya H, Sidana S. Antibody-Based Treatment Approaches in Multiple Myeloma. Curr Hematol Malig Rep. 2021 Apr;16(2):183-191. doi: 10.1007/s11899-021-00624-6. Epub 2021 Mar 17. PMID 33730360
- [Derived] Nooka AK, Weisel K, van de Donk NW, Routledge D, Otero PR, Song K, Quach H, Callander N, Minnema MC, Trudel S, Jackson NA, Ahlers CM, Im E, Cheng S, Smith L, Hareth N, Ferron-Brady G, Brouch M, Montes de Oca R, Paul S, Holkova B, Gupta I, Kremer BE, Richardson P. Belantamab mafodotin in combination with novel agents in relapsed/refractory multiple myeloma: DREAMM-5 study design. Future Oncol. 2021 Jun;17(16):1987-2003. doi: 10.2217/fon-2020-1269. Epub 2021 Mar 8. PMID 33682447

DOCUMENTS (1):
  • Study Protocol (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04126200/Prot_000.pdf